CLINICAL TRIAL: NCT01969266
Title: Open-Label, 2-Period, Sequential Design, Exploratory Pharmacokinetic Study In Healthy Subjects to Assess the Pharmacokinetics and Safety of a Supra-Therapeutic Dose of Ibrutinib Capsule and Solution Formulations Administered With Food
Brief Title: A Pharmacokinetic Study in Healthy Participants to Assess the Pharmacokinetics and Safety of a Supratherapeutic Dose of PCI-32765 (Ibrutinib) Capsule and Solution Formulations Administered With Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR102577; PCI-32765CLL1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-08-19; First posted 2013-10-25 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteer; PCI-32765; PCI 45227; JNJ-54179060; Pharmacokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 (Experimental): PCI-32765 840 mg will be administered as capsule (Treatment A in Period 1) and solution (Treatment B in Period 2) formulations. All participants will receive both treatments with a 7-day washout period between doses.
  Interventions: Drug: Treatment A: PCI-32765; Drug: Treatment B: PCI-32765

INTERVENTIONS:
Drug: Treatment A: PCI-32765 — 840 mg capsule formulation administered by mouth on Day 1
Drug: Treatment B: PCI-32765 — 840 mg solution formulation administered by mouth on Day 1

SUMMARY:
The purpose of this study is to examine the exposure and safety of a supratherapeutic dose of PCI-32765 (ibrutinib) in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known), 2-period, sequential, exploratory study in healthy adult men and women to determine the exposure and safety of a supratherapeutic dose of PCI-32765 (ibrutinib) as a capsule or solution formulation administered with food. Eight participants (including at least 2 women) will be enrolled and receive 2 treatments: PCI-32765 840 mg will be administered as capsule (Treatment A in Period 1) and solution (Treatment B in Period 2) formulations. All participants will receive both treatments with a 7-day washout period between doses. A high-fat breakfast will be provided 2 hours before dosing. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected before dosing and over 72 hours after each dose and safety will be monitored throughout the study. The total duration of the study will be approximately 46 days.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal or surgically sterile
* A sexually active man with a woman of child-bearing potential that has not had a vasectomy must agree to use an adequate contraception method during the study and for 3 months after receiving the last dose of study drug, and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index between 18 and 30 kg/m2 and body weight not less than 50 kg
* Blood pressure (after sitting for 5 minutes) between 90 and 140 mmHg systolic, and no higher than 90 mmHg diastolic
* 12-lead ECG consistent with normal cardiac conduction and function
* Non-smoker

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, history of immune disorders, or any other illness the investigator considers should exclude the participant or could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, PFA 100, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* Use of herbal supplements such as St. John's Wort within 30 days of the first study drug administration
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 2 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening and Day -1 of each treatment period
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water
* A woman that is pregnant, breast-feeding or planning to become pregnant during the study
* A man who plans to father a child while enrolled in the study or within 3 months after the last dose of study drug
* Positive test for human immunodeficiency virus 1 and 2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies
* History of smoking or use of nicotine-containing substances within the previous 2 months, or positive cotinine test at screening
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentrations of ibrutinib and metabolite PCI-45227 | Up to postdose at 72 h
Area under the plasma concentration-time curve of ibrutinib and metabolite PCI-45227 | Up to postdose at 72 h

SECONDARY OUTCOMES:
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States